CLINICAL TRIAL: NCT04719026
Title: PERIODONTAL HEALTH IN PATIENTS ACUTELY ADMITTED FOR MYOCARDIAL INFARCTION: A CASE CONTROL STUDY
Acronym: PEDICAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 203623
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Myocardial Infarction, Acute; Periodontitis
Keywords: myocardial infarction; coronary artery disease; periodontal diseases
MeSH Terms: conditions — Myocardial Infarction; Periodontitis; Coronary Artery Disease; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — subgingival plaque samples, saliva, blood, and in a subgroup of Mi patients (n=10) aspirated intracoronary thrombi and stent deployment ballons used during a primary percutaneous intervention procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients for the case study group will be recruited from those hospitalized for acute myocardial infarction on the Cardiology Ward and Coronary Care Unit at Aberdeen Royal Infirmary. All patients will be diagnosed using current clinical criteria for type-1 myocardial infarction according to the ESC guidelines10 and recruited within 3 days of admission. Recruitment of this arm is now complete.
  Interventions: Other: Full-mouth periodontal examination using computerised Florida probe
- Controls: A control group of dental patients matched for age (±3 years), gender, and risk factors for CAD (hypertension, obesity, diabetes, smoking, hypercholesterolaemia and family history) but with no history of myocardial infarction will be selected at Aberdeen Dental School or from the SHARE register or via the NHS Research Scotland Primary Care Network on an invitation basis. Thr recruitment of this arm of the study is ongoing.
  Interventions: Other: Full-mouth periodontal examination using computerised Florida probe

INTERVENTIONS:
Other: Full-mouth periodontal examination using computerised Florida probe — It is an observational study to investigate the prevalence of periodontitis in cases and controls.

SUMMARY:
Heart attack remains a major cause of death in adult population worldwide and especially within Scotland. A large portion of the general population has an increased risk of suffering from a heart attack because of their genetic make-up, disease profile and lifestyle choices.

Literature suggests that apart from these known risk factors, long-standing inflammation (reaction of tissues to infection or injury) elsewhere in the body may be responsible for heart attacks. It has been suggested that gum disease may be one such condition. If left untreated, gum disease may expose the entire body to a long-term inflammatory burden where inflammatory molecules can disseminate from the gums into the bloodstream and affect various body structures. This study explores the influence of gum disease on the risk of heart attack by comparing the gum health of participants who recently had a heart attack to the gum health of participants with no history of heart problems after accounting for other risk factors. Findings will provide critical information for the design of our forthcoming study to establish the effect of treatment of gum disease on the risk of heart attack, and its cost-effectiveness. Ultimately this research will tackle another risk factor for heart attacks and thus inform enhancement of public health prevention strategies.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is a multifactorial condition leading to most cases of myocardial infarction and results from interaction of genetic, lifestyle and environmental factors. However, as many as 50% of CAD patients lack classical risk factors of CAD suggesting the presence of other contributory mechanisms. Inflammation plays a central role in the initiation and growth of the plaques which form in the arteries (atherosclerosis) and lead to CAD3. As such periodontal disease, an inflammatory process leading to progressive destruction of tooth-supporting structures, has been associated with CAD. In vivo pre-clinical studies have shown that bacteria associated with periodontal disease can exacerbate atherosclerosis 7. Numerous clinical studies have explored the association between periodontal disease and CAD at different follow-up times following episodes of myocardial infarction 8-9. However, there are no reports investigating this association during the acute phase of myocardial infarction. In addition the need for rigorous matching of all known CAD risk factors in case control studies has so far been overseen.

RATIONALE FOR STUDY:

This case-control study aims to compare the health of tooth supporting structures (periodontium) in patients hospitalised for acute myocardial infarction to a control group of patients rigorously matched for known CAD risk factors, age and gender.

ELIGIBILITY:
Inclusion Criteria:

* cases: Patients aged 20-90 admitted with acute myocardial infarction
* controls: Dental patients, aged 20-90, matched to patients in the case study group for age, gender (±7) and risk factors for coronary artery disease (hypertension, obesity, diabetes, smoking, hypercholesterolaemia) but with no history of myocardial infarction)

Exclusion Criteria:

* Severe co-morbidities, Inability to consent, pregnant participants will be excluded, participants with other systemic inflammatory diseases, patients taking antimicrobials or antibiotics in last three years, patients taking medications, such as cyclosporine, calcium channel blockers, phenytoin, immunocompromised patients, patients with malignancies, patinets with type-2 or type-3 hypersensitivities

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients for the case study group will be recruited from those hospitalized for acute myocardial infarction on the Cardiology Ward and Coronary Care Unit at Aberdeen Royal Infirmary.
  A control group of dental patients matched for age (±7 years), gender, and risk factors for CAD (hypertension, obesity, diabetes, smoking, hypercholesterolemia, and family history) but with no history of myocardial infarction will be selected at Aberdeen Dental School or from the SHARE register or via the NHS Research Scotland Primary Care Network
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2018-02-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of periodontitis | Single point examination
  Our primary objective is the description of periodontal health in patients admitted with acute myocardial infarction compared to matched controls

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Karolin Hijazi, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Joshi C, Mezincescu A, Gunasekara M, Rudd A, Botchorichvili H, Sabir S, Dospinescu C, Noman A, Hogg D, Cherukara G, McLernon D, Hijazi K, Dawson D. Myocardial infarction risk is increased by periodontal pathobionts: a cross-sectional study. Sci Rep. 2022 Nov 3;12(1):18608. doi: 10.1038/s41598-022-19154-z. PMID 36329042